CLINICAL TRIAL: NCT01608334
Title: Comparison of Intrathecal Fentanyl or Sufentanil in 1 mg Bupivacaine Spinal Anesthesia for TURP in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2011-0162
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Adequate Anesthesia With Unimpaired Motor Strength
MeSH Terms: interventions — Fentanyl; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Experimental): Fentanyl
  Interventions: Drug: Fentanyl
- Group B (Active Comparator): Sufentanil
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Fentanyl — 1mg 0.5% bupivacaine + fentanyl 20 mcg + 1.8 ml glucose ( total 2.4-ml) VS 1mg 0.5% bupivacaine + sufentanil 5 mcg + 2.1ml glucose (total 2.4-ml) intrathecally.
  Arms: group A
Drug: Sufentanil — 1mg 0.5% bupivacaine + fentanyl 20 mcg + 1.8 ml glucose ( total 2.4-ml) VS 1mg 0.5% bupivacaine + sufentanil 5 mcg + 2.1ml glucose (total 2.4-ml) intrathecally.
  Arms: Group B

SUMMARY:
Adequate sensory block for surgical procedure without side effects and immediate mobilization after surgery are desirable anesthetic technique in various surgeries. Considering the sensory innervations to the prostate, a sensory block up to L1 - T12 is adequate to the TURP. Low-dose intrathecal local anesthetics may meet these criteria, but occasional lack of sufficient sensory block could be troublesome. In this randomized study, the investigators evaluated the spinal anesthetic characteristics following intrathecal administration of bupivacaine 1 mg with fentanyl or sufentanil in elderly patients undergoing TURP.

ELIGIBILITY:
Inclusion Criteria:

* age over 65 ~ under 85yrears old
* male
* elderly patients undergoing TURP
* only spinal anesthesia
* patients consent about this study

Exclusion Criteria:

* spine surgery History
* coagulopathy
* impaired communication
* impaired orientation
* DM complication neuropathy
* BMI > 30 -> overweight patients.

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
time to achieve peak sensory block without unimpaired motor strength | 2 minites after injection intrathecally start
  peak sensory & sympathetic block level, time to peak sensory & sympathetic block level, motor block level at peak sensory & sympathetic block level, lowest BP and HR during spinal anestheisa, frequency of painkiller

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea